CLINICAL TRIAL: NCT01158274
Title: A Phase 1 Study of RO4929097 (NSC749225) in Combination With Capecitabine in Refractory Solid Tumors
Brief Title: RO4929097 and Capecitabine in Treating Patients With Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02918; NCI-2012-02918 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000680610; CO09907 (Other: University of Wisconsin Hospital and Clinics); 8515 (Other: CTEP); U01CA062491 (NIH); U01CA132123 (NIH); P30CA014520 (NIH)
Record Dates: First submitted 2010-07-07; First posted 2010-07-08 (Estimated); Last update posted 2014-11-07 (Estimated); Status verified 2014-06

CONDITIONS: Adult Grade III Lymphomatoid Granulomatosis; Adult Nasal Type Extranodal NK/T-cell Lymphoma; AIDS-related Diffuse Large Cell Lymphoma; AIDS-related Diffuse Mixed Cell Lymphoma; AIDS-related Diffuse Small Cleaved Cell Lymphoma; AIDS-related Immunoblastic Large Cell Lymphoma; AIDS-related Lymphoblastic Lymphoma; AIDS-related Peripheral/Systemic Lymphoma; AIDS-related Primary CNS Lymphoma; AIDS-related Small Noncleaved Cell Lymphoma; Anaplastic Large Cell Lymphoma; Angioimmunoblastic T-cell Lymphoma; Cutaneous B-cell Non-Hodgkin Lymphoma; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; HER2-negative Breast Cancer; HIV-associated Hodgkin Lymphoma; Intraocular Lymphoma; Male Breast Cancer; Nodal Marginal Zone B-cell Lymphoma; Post-transplant Lymphoproliferative Disorder; Primary Central Nervous System Hodgkin Lymphoma; Primary Central Nervous System Non-Hodgkin Lymphoma; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Grade III Lymphomatoid Granulomatosis; Recurrent Adult Hodgkin Lymphoma; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Adult T-cell Leukemia/Lymphoma; Recurrent Breast Cancer; Recurrent Colon Cancer; Recurrent Cutaneous T-cell Non-Hodgkin Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Mycosis Fungoides/Sezary Syndrome; Recurrent Rectal Cancer; Recurrent Small Lymphocytic Lymphoma; Small Intestine Lymphoma; Splenic Marginal Zone Lymphoma; Stage III Adult Burkitt Lymphoma; Stage III Adult Diffuse Large Cell Lymphoma; Stage III Adult Diffuse Mixed Cell Lymphoma; Stage III Adult Diffuse Small Cleaved Cell Lymphoma; Stage III Adult Hodgkin Lymphoma; Stage III Adult Immunoblastic Large Cell Lymphoma; Stage III Adult Lymphoblastic Lymphoma; Stage III Adult T-cell Leukemia/Lymphoma; Stage III Colon Cancer; Stage III Cutaneous T-cell Non-Hodgkin Lymphoma; Stage III Grade 1 Follicular Lymphoma; Stage III Grade 2 Follicular Lymphoma; Stage III Grade 3 Follicular Lymphoma; Stage III Mantle Cell Lymphoma; Stage III Marginal Zone Lymphoma; Stage III Mycosis Fungoides/Sezary Syndrome; Stage III Rectal Cancer; Stage III Small Lymphocytic Lymphoma; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer; Stage IV Adult Burkitt Lymphoma; Stage IV Adult Diffuse Large Cell Lymphoma; Stage IV Adult Diffuse Mixed Cell Lymphoma; Stage IV Adult Diffuse Small Cleaved Cell Lymphoma; Stage IV Adult Hodgkin Lymphoma; Stage IV Adult Immunoblastic Large Cell Lymphoma; Stage IV Adult Lymphoblastic Lymphoma; Stage IV Adult T-cell Leukemia/Lymphoma; Stage IV Breast Cancer; Stage IV Colon Cancer; Stage IV Cutaneous T-cell Non-Hodgkin Lymphoma; Stage IV Grade 1 Follicular Lymphoma; Stage IV Grade 2 Follicular Lymphoma; Stage IV Grade 3 Follicular Lymphoma; Stage IV Mantle Cell Lymphoma; Stage IV Marginal Zone Lymphoma; Stage IV Mycosis Fungoides/Sezary Syndrome; Stage IV Rectal Cancer; Stage IV Small Lymphocytic Lymphoma; Unspecified Adult Solid Tumor, Protocol Specific; Waldenström Macroglobulinemia
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Intraocular Lymphoma; Breast Neoplasms, Male; Lymphoma, B-Cell, Marginal Zone; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Breast Neoplasms; Colonic Neoplasms; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Rectal Neoplasms; Leukemia, Lymphocytic, Chronic, B-Cell; Waldenstrom Macroglobulinemia | interventions — 2,2-dimethyl-N-(6-oxo-6,7-dihydro-5H-dibenzo(b,d)azepin-7-yl)-N'-(2,2,3,3,3-pentafluoropropyl)malonamide; Capecitabine

ARMS (1):
- Treatment (Experimental): Patients receive oral gamma-secretase inhibitor RO4929097 once daily on days 1-3, 8-10, and 15-17 and oral capecitabine twice daily on days 1-14. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: gamma-secretase/Notch signalling pathway inhibitor RO4929097; Drug: capecitabine; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: gamma-secretase/Notch signalling pathway inhibitor RO4929097 — Given orally
  Other Names: R4733; RO4929097
Drug: capecitabine — Given orally
  Other Names: CAPE; Ro 09-1978/000; Xeloda
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I clinical trial is studying the side effects and best dose of RO4929097 when given together with capecitabine in treating patients with refractory solid tumors. RO4929097 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving RO4929097 together with chemotherapy may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of RO4929097 and capecitabine administered in subjects with advanced solid tumors. (Part 1) II. To describe the dose-limiting toxicities (DLTs) of combined RO492097 and capecitabine. (Part 1) III. To determine the safety of RO4929097 and capecitabine administered in combination. (Part 1) IV. To determine the safety of RO4929097 and capecitabine in subjects with metastatic CRC. (Part 2a) V. To evaluate the safety of RO4929097 and capecitabine in combination for subjects with HER2/neu negative MBC. (Part 2b)

SECONDARY OBJECTIVES:

I. To determine the clinical activity of RO4929097 and capecitabine administered in combination to subjects with advanced solid tumors. (Parts 1, 2a, and 2b) II. To evaluate the changes in the expression of Notch1 signaling pathway members and downstream targets of Notch by PCR including HEs1, 3 and 5; Hey 1 and 2 after treatment with RO4929097 at the MTD expansion cohorts. (Parts 1, 2a, and 2b) III. To determine the pharmacokinetic and pharmacogenomic profiles of the combination of RO4929097 and capecitabine. (Parts 1, 2a, and 2b) IV. To determine the progression-free survival (PFS) of RO4929097 and capecitabine when administered at the MTD level in patients with metastatic colorectal cancer (CRC) and a history of 1 or 2 prior therapies. (Part 2a) V. To determine the response and overall survival (OS) rates following RO4929097 and capecitabine administration at the MTD level in subjects with metastatic CRC. (Part 2a) VI. To determine the overall response rate (ORR) of RO4929097 and capecitabine when administered at the MTD level to subjects when administered first or second line for HER2/neu negative metastatic breast cancer (MBC). (Part 2b) V. To determine the progression-free and overall survival rates following RO4929097 and capecitabine administration at the MTD level in subjects with HER2/neu negative MBC. (Part 2b)

OUTLINE: This is a multicenter, dose-escalation study of gamma-secretase inhibitor RO4929097.

Patients receive oral gamma-secretase inhibitor RO4929097 once daily on days 1-3, 8-10, and 15-17 and oral capecitabine twice daily on days 1-14. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Patients may undergo tumor biopsy before and after treatment for biomarker analysis and blood sample collection periodically for pharmacokinetic and pharmacogenomic studies.

After completion of study treatment, patients are followed up for 30 days (Part 1) or every 3 months (Parts 2a and 2b).

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed advanced or metastatic solid tumor; patients with lymphoma will be eligible
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 20 mm with conventional techniques or as >= 10 mm with spiral CT scan
* Patients must be at least 4 weeks since prior chemotherapy, 6 weeks if the last regimen included BCNU or mitomycin C; prior radiation is allowed as long as the radiation was completed 4 weeks prior to study treatment and no more than 35% of marrow irradiated
* Life expectancy of greater than 3 months
* ECOG performance status =< 2 (Karnofsky >= 60%)
* Hemoglobin >= 9 g/dL
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin within normal institutional limits
* AST (SGOT)/ALT (SGPT) =< 2.5 X institutional upper limit of normal
* Creatinine within normal institutional limits OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal; a 24 hour urine collection and creatinine clearance can be measured if indicated
* Treated, stable brain metastases are allowed; patients must be four weeks from radiation with stable brain imaging and off any medications used to treat brain metastases, excepting those anti-epileptics not metabolized by cytochrome P450
* Women of childbearing potential and men must use two forms of contraception (i.e., barrier contraception and one other method of contraception) at least 4 weeks prior to study entry, for the duration of study participation, and for at least 12 months post-treatment; should a woman become pregnant or suspect she is pregnant while she or her partner are participating in this study and for 12 months after study participation, the patient should inform the treating physician immediately
* Women of childbearing potential are required to have a negative serum pregnancy test (with a sensitivity of at least 25 mIU/mL) within 10-14 days and within 24 hours prior to the first dose of RO4929097 (serum or urine); a pregnancy test (serum or urine) will be administered every 4 weeks if their menstrual cycles are regular or every 2 weeks if their cycles are irregular while on study within the 24-hour period prior to the administration of RO4929097; a positive urine test must be confirmed by a serum pregnancy test; prior to dispensing RO4929097, the investigator must confirm and document the patient's use of two contraceptive methods, dates of negative pregnancy test, and confirm the patient's understanding of the teratogenic potential of RO4929097
* Female patients of childbearing potential are defined as follows:

  * Patients with regular menses
  * Patients, after menarche with amenorrhea, irregular cycles, or using a contraceptive method that precludes withdrawal bleeding
  * Women who have had tubal ligation
* Female patients may be considered NOT to be of childbearing potential for the following reasons:

  * The patient has undergone total abdominal hysterectomy with bilateral salpingo-oophorectomy or bilateral oophorectomy
  * The patient is medically confirmed to be menopausal (no menstrual period) for 24 consecutive months
  * Pre-pubertal females. The parent or guardian of young female patients who have not yet started menstruation should verify that menstruation has not begun. If a young female patient reaches menarche during the study, then she is to be considered as a woman of childbearing potential from that time forward
* Patients must demonstrate an ability to understand and the willingness to sign a written informed consent document
* Preclinical studies indicate that RO4929097 is a substrate of CYP3A4 and inducer of CYP3A4 enzyme activity; caution should be exercised when dosing RO4929097 concurrently with CYP3A4 substrates, inducers, and/or inhibitors; furthermore, patients who are taking concurrent medications that are strong inducers/inhibitors or substrates of CYP3A4 should be switched to alternative medications to minimize any potential risk; if such patients cannot be switched to alternative medications, they will be ineligible to participate in this study
* PART 2A (MTD EXPANSION COLORECTAL CANCER):
* For this cohort patients must have histologically or cytologically documented advanced or metastatic colorectal cancer; patients must have had at least one prior chemotherapy regimen for their disease but no more than 2
* All 5 patients in this cohort must be willing and able to have tumor biopsies performed as part of the correlative studies associated with this trial
* PART 2B (MTD EXPANSION BREAST CANCER):
* For this cohort, patients must have histologically or cytologically documented advanced or metastatic breast cancer
* Patient must be HER2/neu negative; HER2 negative will be defined as HER2 neither over-expressed or amplified; HER2 will be considered NOT over-expressed if the tumor stains as 0 or 1+ for HER2 by immunohistochemistry (IHC); if the IHC for HER2 is 2+, fluorescence in-site hybridization (FISH) ratio must be less than 2 to be considered NOT amplified; any tumor for which only FISH was performed must have a ratio of less than 2 to be considered NOT amplified
* All 5 patients in this breast cancer cohort must be willing and able to have tumor biopsies performed as part of the correlative studies associated with this trial

Exclusion Criteria:

* Patients may not be receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to RO4929097 or capecitabine
* Patients taking medications with narrow therapeutic indices that are metabolized by cytochrome P450 (CYP450), including warfarin sodium (Coumadin®) are ineligible
* Patients with malabsorption syndrome or other condition that would interfere with intestinal absorption; patients must be able to swallow tablets
* Patients who are serologically positive for Hepatitis A, B or C, or have a history of liver disease, other forms of hepatitis or cirrhosis are ineligible
* Patients with uncontrolled hypocalcemia, hypomagnesemia, hyponatremia, hypophosphatemia or hypokalemia defined as less than the lower limit of normal for the institution, despite adequate electrolyte supplementation are excluded from this study; note: it is acceptable to use corrected calcium when interpreting calcium levels
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, and a history of torsades de pointes or other significant cardiac arrhythmia other than chronic, stable atrial fibrillation, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued
* HIV-positive patients, who are not on anti-retroviral therapy but have CD4 cells less than 200, should be excluded; HIV-positive patients are eligible if they are on HAART (highly active anti-retroviral therapy) which are not CYP3A4 substrates, inducers and/or inhibitors and meet all other criteria
* Cardiovascular: baseline QTcF > 450 msec
* Patients with known dihydropyrimidine dehydrogenase (DPD) deficiency enzyme are excluded
* Patients who have not recovered to < CTCAE grade 2 toxicities related to prior therapy are not eligible to participate in this study
* A requirement for antiarrhythmics or other medications known to prolong QTc
* PART2B (MTD EXPANSION BREAST CANCER):
* Patients may not have had more than 1 prior cytotoxic chemotherapy for metastatic disease; prior endocrine or immunotherapy regimens for metastatic disease will not be counted as cytotoxic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-06; Primary Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
MTD of RO4929097 and capecitabine, defined as that dose level at which less than one-third of patients experience a dose-limiting toxicity (DLT) graded according to NCI CTCAE version 4.0 (Part 1) | Up to 21 days
Incidence of adverse events graded according to NCI CTCAE version 4.0 (Part 1) | Up to 30 days after completion of study treatment
  Possible adverse events will be reported in tabular format. To determine the severity of the reaction for adverse event reporting, the NCI CTCAE version 4.0 will be used.
Incidence of adverse events graded according to NCI CTCAE version 4.0 (Parts 2a and 2b) | Up to 24 months
  Possible adverse events will be reported in tabular format. To determine the severity of the reaction for adverse event reporting, the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be used.

SECONDARY OUTCOMES:
Confirmed anti-tumor response rate validated by the RECIST (Part 1) | Up to 30 days after completion of study treatment
  Responses will be summarized using descriptive statistics presented in tabular format. Furthermore, two-sided 95% confidence intervals for the proportions of subjects with a confirmed anti-tumor response will be computed, while adjusting for multiplicity.
Changes in the expression of Notch1 signaling pathway members (Part 1) | From baseline to 30 days after completion of study treatment
  Relative and absolute changes will be calculated for each patient and results will be summarized by means and standard deviations. Paired t-tests will be used to compare baseline and post-study values in expression levels.
Pharmacokinetics of the combination of RO4929097 and capecitabine, including Cmax, Tmax, AUC, t1/2, and CL (Part 1) | Baseline on day 1 of course 1; baseline and 1, 2, 3, 4, 8, 12, 16, and 24 hours on days 3 and 10 of course 1; and baseline on day 1 of all subsequent courses
  PK parameters will be summarized by using means, standard deviations and ranges. PK parameters between patients with a response (partial or complete) will be compared to PK parameters of patients with no response using a nonparametric Wilcoxon Rank Sum test.
PFS (Parts 2a and 2b) | Up to 24 months
  Presented in a tabular format.
OS (Part 2a and 2b) | Number of days from the day of first RO4929097 and capecitabine administration to the patient's death, assessed up to 24 months
  Presented in a tabular format.
Overall response rate (Parts 2a and 2b) | Up to 24 months
  Confirmed anti-tumor response rate will be validated by RECIST. Responses will be summarized using descriptive statistics presented in tabular format.

CONTACTS AND LOCATIONS:
Overall Officials: Noelle LoConte, Principal Investigator — University of Wisconsin, Madison
Locations (2):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States
- University Health Network-Princess Margaret Hospital, Toronto, Ontario, Canada